CLINICAL TRIAL: NCT00871481
Title: Laboratory-Treated T Cells and Ipilimumab in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2225.00; NCI-2010-00108 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K12CA076930 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Cyclophosphamide; Biopsy; aldesleukin; Interleukin-2; Immunohistochemistry; Polymerase Chain Reaction; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (laboratory-treated T cells and ipilimumab) (Experimental): Patients receive cyclophosphamide IV on day -2, therapeutic cytotoxic T lymphocytes IV over 30-60 minutes on day 0, low-dose aldesleukin SC BID on days 0-13, and ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ipilimumab; Drug: cyclophosphamide; Procedure: biopsy; Biological: aldesleukin; Other: immunohistochemistry staining method; Genetic: polymerase chain reaction; Other: immunoenzyme technique; Biological: therapeutic cytotoxic T lymphocytes

INTERVENTIONS:
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Biological: therapeutic cytotoxic T lymphocytes — Given IV
  Other Names: therapeutic CTLs

SUMMARY:
This phase I/II trial is studying the side effects of giving laboratory-treated T cells and ipilimumab together to see how well they work in treating patients with metastatic melanoma. Treating a patient's T cells in the laboratory may help the T cells kill more tumor cells when they are put back in the body. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving laboratory-treated T cells together with ipilimumab may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and efficacy of adoptively transferred cytotoxic lymphocytes (CTL) targeting melanoma tumors combined with anti-CTLA4.

II. Evaluate the influence of anti-CTLA4 (ipilimumab) on the duration of in vivo persistence and anti-tumor efficacy achieved following adoptive transfer of antigen-specific CTL.

SECONDARY OBJECTIVES:

I. Evaluate the influence of anti-CTLA4 on the induction of T cells to non-targeted tumor-associated antigens (antigen-spreading) following adoptive transfer antigen-specific CTL, and the correlation of these responses with clinical outcome.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) on day -2, therapeutic cytotoxic T lymphocytes IV over 30-60 minutes on day 0, low-dose aldesleukin subcutaneously (SC) twice daily (BID) on days 0-13, and ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic documentation of melanoma concurrent with the diagnosis of metastatic disease
* Expression of human leukocyte antigen (HLA)-A2
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-1
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized; suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion, and at least 8 weeks after the study drug is stopped; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal
* Men must be willing and able to use an acceptable method of birth control, for at least 3 months after completion of the study, if their sexual partners are WOCBP
* Willing and able to give informed consent
* Adequate venous access-consider peripherally inserted central catheter (PICC) or central line
* Bi-dimensionally measurable disease by palpation on clinical exam, or radiographic imaging (X-ray, computed tomography [CT] scan)
* At least 4 weeks must have elapsed since the last chemotherapy, radiotherapy or major surgery; at least 6 weeks for nitrosoureas, mitomycin C and liposomal doxorubicin; if started before T-cell administration, Ipilimumab infusions must be least 21 days apart
* Toxicity related to prior therapy must either have returned to =< grade 1, baseline, or been deemed irreversible
* Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after study drug is stopped

Exclusion Criteria:

* Patients with active infections or oral temperature > 38.2 C within 72 hours prior to planned leukapheresis; the procedure may be deferred
* Patients with hematocrit (Hct) < 30%, white blood cells (WBC) < 2500/uL and platelets < 50,000 immediately prior to leukapheresis; the procedure may be deferred
* Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix
* White blood cell count (WBC) < 2000/uL
* Hematocrit (Hct) < 24% or hemoglobin (Hb) < 8 g/dL
* Absolute neutrophile count (ANC) < 1000
* Platelets < 50,000
* Creatinine > 3.0 x upper limit normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2.5 x ULN
* Bilirubin > 3 x ULN
* Pregnant women, nursing mothers, men or women of reproductive ability who are unwilling to use effective contraception; women of childbearing potential with a positive pregnancy test within 3 days prior to entry
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 2.0 L or diffusion capacity of carbon monoxide (DLco) (corr for Hgb) < 50% will be excluded
* Significant cardiovascular abnormalities as defined by any one of the following:

  * Congestive heart failure
  * Clinically significant hypotension
  * Symptoms of coronary artery disease
  * Presence of cardiac arrhythmias on electrocardiogram (EKG) requiring drug therapy
  * Ejection fraction < 50 % (echocardiogram or multi gated acquisition [MUGA] scan)
* Active and untreated central nervous system (CNS) metastasis (including metastasis identified during screening magnetic resonance imaging [MRI] or contrast CT)
* Autoimmune disease: Patients with a history of Inflammatory Bowel Disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the Investigator to be unacceptable
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Positive screening tests for human immunodeficiency virus (HIV), hepatitis (Hep) B, and Hep C; if positive results are not indicative of true active or chronic infection, the patient can be treated
* Steroids are not permitted 3 days prior to T cell infusion and concurrently during therapy
* No prisoners or children will be enrolled on this study
* Any non-oncology vaccine therapy used for the prevention of infectious disease within 1 month before or after any ipilimumab dose
* Patients may not be on any other treatments for their cancer aside from those included in the protocol; patients may not undergo another form of treatment concurrently with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Numeric frequency and functional persistence of transferred CTL | Up to 6 months post-infusion
  Determined using peptide major histocompatibility complex (MHC)-tetramer analysis or specific CDR3 T-cell-receptor (TCR) quantitative polymerase chain reaction (PCR) of transferred CTL if necessary. The function of transferred CTL will be determined by intracellular cytokine staining of tetramer+ CD8+ cells following in vitro stimulation.
Toxicity assessment of study treatment, assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 | Up to 6 months post-infusion

SECONDARY OUTCOMES:
Responses to non-targeted T cell antigens | Up to 1 year following T cell infusion and/or at the time of observed partial or complete clinical response
  Blood samples taken will be analyzed for the induction of non-targeted T cell responses. Two approaches will be used: tetramer analysis and enzyme-linked immunosorbent spot (ELISPOT) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Aude Chapuis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Chapuis AG, Roberts IM, Thompson JA, Margolin KA, Bhatia S, Lee SM, Sloan HL, Lai IP, Farrar EA, Wagener F, Shibuya KC, Cao J, Wolchok JD, Greenberg PD, Yee C. T-Cell Therapy Using Interleukin-21-Primed Cytotoxic T-Cell Lymphocytes Combined With Cytotoxic T-Cell Lymphocyte Antigen-4 Blockade Results in Long-Term Cell Persistence and Durable Tumor Regression. J Clin Oncol. 2016 Nov 1;34(31):3787-3795. doi: 10.1200/JCO.2015.65.5142. PMID 27269940